CLINICAL TRIAL: NCT05950633
Title: Evaluating a Novel Active Recovery Program in the Immediate Postoperative Period Following Pelvic Reconstructive Surgery: A Randomized Control Trial
Brief Title: Postoperative Active Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sara Cichowski, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 25625
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Participants will receive standard postoperative instructions only
  Interventions: Other: Standard of Care
- Active Recovery (Active Comparator): Participants will receive active recovery instructions with specific walking goals, abdominal strengthening exercises, and pelvic floor exercises
  Interventions: Other: Active Recovery

INTERVENTIONS:
Other: Standard of Care — Participants will receive standard of care postoperative instructions
  Arms: Standard of Care
Other: Active Recovery — Participants will receive instructions to increase their fitness to walking at least 30 minutes a day for 5 days a week following surgery and abdominal and pelvic floor exercises will focus on abdominal wall strengthening and abdominal pressure management, urinary urgency and retention, bowel and constipation management
  Arms: Active Recovery

SUMMARY:
This is a study evaluating a novel active recovery program in the immediate postoperative period following pelvic reconstructive surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing usual care postoperative restrictions and a novel new active recovery program to look at differences in pelvic floor function, patient quality of life, and mental health in between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 89
2. Undergoing minimally invasive apical prolapse reconstructive procedure at OHSU. This includes laparoscopic and robotic-assisted sacrocolpopexy, laparoscopic and vaginal uterosacral ligament suspension, and vaginal sacrospinous ligament fixation. We will include patients undergoing concomitant procedures such as hysterectomy and incontinence procedures.
3. Have access to reliable email for communication and questionnaires.

Exclusion Criteria:

1. Unable to consent
2. Unable to read and complete questionnaires in English
3. Unable to sustain 30 minutes of moderate walking/activity at baseline (self-reported)
4. Use a mobility assistance device such as a walker/cane at baseline
5. Balance or stability problems
6. Patients on chronic opioids

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the Pelvic Floor Distress Inventory-20 (PFDI-20) | Baseline to 12 weeks post-surgery
  The change in the Pelvic Floor Distress Inventory-20 (PFDI-20) between arms from baseline to 12 weeks post-surgery. Participants will be asked to rate how much symptoms bother them from 0 (not at all) to 4 (quite a bit)
Change in the Short Form Health Survey (SF-36) | Baseline to 12 weeks
  The change in the Short Form Health Survey (SF-36) between arms from baseline to 12 weeks post-surgery. Participants will be asked to rate their overall health. Scores can range from 0 to 100
Change in the Patient Health Questionnaire (PHQ-9) | Baseline to 12 weeks post-surgery
  The change in the Patient Health Questionnaire (PHQ-9) between arms from baseline to 12 weeks post-surgery. Participants will be asked to rate how frequently problems have bothered them from 0 (not at all) to 4 (nearly every day)
Change in the Patient Global Impression of Improvement (PGI-I) | Baseline to 12 weeks post-surgery
  The change in the Patient Global Impressions of Improvement (PGI-I) between arms from baseline to 12 weeks post-surgery. Participants will be asked to rate their symptoms from 1 (very much better) to 7 (very much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cichowski, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States